CLINICAL TRIAL: NCT06002451
Title: The Effect of Web-based Preconceptional Care and Counseling on Risk Awareness and Healthy Lifestyle Behavior in Women
Brief Title: Web-based Preconceptional Care and Counseling, Risk Awareness, Healthy Lifestyle Behavior
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Öznur HASDEMİR, midwife, Cumhuriyet University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: CUMHURIYET UNIVERSITY HASDEMIR
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Web
Keywords: Risk Awareness; Web-based; Preconceptional Care; Preconceptional Counselling; Innovation; Midwifery; Training; Healthy Lifestyle
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WEB-BASED PRECONCEPTİONAL CARE AND COUNSELİNG (Experimental): At the beginning of the study, Pre-test Forms were applied and data were obtained.A total of 9 Module Trainings for PC and maintenance were given over the Web Base for 2 weeks. While the trainings were continuing, the modules were monitored from the Admin Panel and reminder messages were sent to the people who did not watch the modules regularly. During the training, PD and care services were provided via the communication. At the end of the 10th week, the post-test forms were applied and the data were obtained. that they can reach 24/7 for a total of 10 weeks, 2 weeks and the following 8 weeks.
  Interventions: Behavioral: WEB-BASED PRECONCEPTİONAL CARE AND COUNSELİNG
- CONTROL (No Intervention): Pre-test Forms were applied and data were obtained.No attempt has been made. This group received routine training and follow-ups at the family health center and premarital counseling unit.At the end of the 10th week, the post-test forms were applied and the data were obtained.

INTERVENTIONS:
Behavioral: WEB-BASED PRECONCEPTİONAL CARE AND COUNSELİNG — A web-based preconceptional care and consultancy training platform has been developed. In line with the literature, a comprehensive preconceptional care and counseling training content was prepared for women between the ages of 18-49. Web-based training consists of a total of 9 modules.The videos created for uploading to the website were shot in a professional studio environment with professional equipment.Each video was shot and recorded by dividing the training content according to its subsections, with an average of at least 6 minutes and a maximum of 16 minutes. Each of the module videos is based on giving the main messages in line with the purpose and objectives of the presentation.women were allowed to watch all the videos within 2 weeks. A dialog box is opened on the website where women can communicate with their midwives 24/7. During and after the training, preconceptional care and counseling training was given in this area for a total of 10 weeks.
  Arms: WEB-BASED PRECONCEPTİONAL CARE AND COUNSELİNG

SUMMARY:
Preconceptional (pre-pregnancy) care; It is a primary care preventive health service that aims to prepare individuals for pregnancy, to maintain and result in a healthy pregnancy process, and thus to contribute to the formation of new generations from healthier individuals. The purpose of preconceptional care; identifying the risk factors present in the woman is to eliminate or reduce the adverse effects of these risk factors in the pregnancy process, improve health, improve mother and child health in the short and long term. Preconception counseling (PC), on the other hand, is to provide training on the best way to achieve a healthy pregnancy by addressing women's existing health problems and modifiable risk factors. When performing PC and care, it is necessary to maintain a system based on evidence and to assess women's holistic and create risk awareness. The creation of risk awareness in women should begin with the determination of the risk factors present before pregnancy. It is also very important to identify pre-pregnancy risk factors and to provide healthy lifestyle behaviors. Today, web-based training is known to be used to adapt individuals to new situations and to improve the health of individuals, to improve positive behavior changes.This research was conducted to determine the effect of web-based preconceptional care and counseling on risk awareness and healthy lifestyle behavior in women.

DETAILED DESCRIPTION:
Planning fertility with evidence-based management while providing preconceptional care and counseling; advanced maternal and paternal age; family history, genetic history and diseases; physical activity, body mass index; nutrition; vaccination; sexually transmitted infections; chronic diseases; drugs ;harmful habits and exposure; Psychosocial sub-dimensions of women should be evaluated holistically and risk awareness should be created.As a matter of fact, creating risk awareness in women should start with the identification of risk factors that exist before pregnancy. It is possible to gain healthy lifestyle behaviors with the determination of these risk factors and taking the necessary precautions.Studies have shown that preconception care and counseling services provide cost-effectiveness while improving maternal and child health; It is emphasized that health institutions that are inadequate in providing this service should develop strategies to encourage preconceptional care and counseling at the community level, especially for women.Recommendations of reputable organizations such as CDC, ACOG, WHO; It has been concluded that preconceptional care and counseling services should be expanded more effectively and quickly in line with the results and recommendations of the researches; It is thought that this widespread effect can be achieved by using the internet and web-based trainings, which are a part of our lives.It is reported in the literature that web-based trainings are seen as an appropriate intervention area in reaching women of childbearing age who need preconceptional care and counseling.Although there are studies in the world that web-based PC and care services are provided and that they affect health positively; No studies on web-based PC and maintenance services have been found in our country.The results obtained from this study; establishing a comprehensive evidence-based standard PC and maintenance program; improving risk awareness and healthy lifestyle behaviors of women of childbearing age; It is thought that it will lead to the encouragement of the use of modern technology areas in the field of PC and care services, to the development of all health personnel, especially midwives, who want to provide comprehensive services in this field, to use web-based PC and maintenance program in field applications, and to contribute to the midwifery literature in the planning of advanced studies. .

ELIGIBILITY:
Inclusion Criteria:

* Literate,
* Between the ages of 18-49, who are of childbearing age,
* Not pregnant,
* Not receiving preconceptional care and consultancy services,
* Does not have a disorder based on a psychiatric/psychological diagnosis,
* No diagnosis of menopause,
* Internet access,
* Using at least one computer-tablet-smartphone,
* Communicable and language-free

Exclusion Criteria:

* Those who do not agree to participate in the research,
* under 18 years old and over 49 years old,
* pregnant,
* Receiving preconceptional care and counseling before,
* illiterate,
* No internet access,
* Not having at least one computer-tablet-smartphone,
* Having a disorder based on a psychiatric/psychological diagnosis,
* Diagnosed with menopause,
* Having communication and language problems.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — It covers women of childbearing age between the ages of 18-49.
Enrollment: 84 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2023-07-09 (Actual)

PRIMARY OUTCOMES:
risk awareness in women | 10 week
  The research is an experimentally planned randomized controlled trial. The sample of the study consists of women between the ages of 18-49 who are in the reproductive age. Women's risk awareness was evaluated with the Preconceptional period risk awareness scale, which was developed in line with preconceptional care and counseling. All statements of the scale, which consists of 37 items in total, are positive. The lowest score obtained from the scale is 37, and the highest score is 185. The scale has no breakpoints. The total score of the scale determines the preconceptional period risk awareness score. As the scores obtained from the scale increase, women's preconceptional period risk awareness levels increase. The Cronbach Alpha coefficient of the scale is 0.90 and it has a high degree of reliability.

SECONDARY OUTCOMES:
Healthy lifestyle behaviors of women | 10 week
  The research is an experimentally planned randomized controlled trial. The sample of the study consists of women between the ages of 18-49 who are in the reproductive age. Health-promoting behaviors of women in relation to a healthy lifestyle were evaluated with the Healthy Lifestyle Behaviors Scale-II. The lowest score for the whole scale is 52, and the highest score is 208. The scale has no breakpoints. The total score of the scale determines the healthy lifestyle behaviors score. The Cronbach Alpha coefficient of the scale is 0.92 and it has a high degree of reliability.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Burcu YURTSAL, Assoc. Prof., Study Director — Sivas Cumhuriyet University, Faculty of Health Sciences, Department of Midwifery, Sivas; Öznur HASDEMİR, PhD, Principal Investigator — PROVINCIAL HEALTH DIRECTORATE, PUBLIC HEALTH SERVICES, SİVAS
Locations (1):
- Community health center and family health centers affiliated to Sivas Provincial Health Directorate, Sivas, Center/ Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The women were informed about the research subject and purpose, and their written and verbal informed consent was obtained. The study was conducted in accordance with the Principles of the Declaration of Helsinki.